CLINICAL TRIAL: NCT03509220
Title: A Prospective, Randomized, Parallel, Multi-center, Phase 3 Trial to Evaluate Safety and Efficacy of PBK-1701TC
Brief Title: Safety and Efficacy of PBK-1701TC for Bowel Cleansing Before Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmbio Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PBK-1701TC_P3
Record Dates: First submitted 2018-04-11; First posted 2018-04-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Colonic Diseases; Intestinal Disease; Gastrointestinal Disease; Digestive System Disease
Keywords: Colonoscopy; PBK-1701TC; Bowel cleansing
MeSH Terms: conditions — Colonic Diseases; Intestinal Diseases; Gastrointestinal Diseases; Digestive System Diseases | interventions — pbk-1701TC

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PBK-1701TC (Experimental): 2-Day Split-Dosing Regimen
  Interventions: Drug: PBK-1701TC
- Standard oral preparation (Active Comparator): 2-Day Split-Dosing Regimen
  Interventions: Drug: Standard oral preparation

INTERVENTIONS:
Drug: PBK-1701TC — The subject will receive PBK-1701TC for colonoscopy.
  Arms: PBK-1701TC
Drug: Standard oral preparation — The subject will receive the standard oral preparation for colonoscopy
  Arms: Standard oral preparation

SUMMARY:
This study evaluates the efficacy, safety and tolerability of PBK-1701TC for bowel cleansing before colonoscopy. Half the participants will receive PBK-1701TC and while the other will receive standard oral preparation.

DETAILED DESCRIPTION:
This study is a prospective, randomized, single-blinded, parallel, 2-treatment, multi-center clinical trial. A total of 224 subjects will participate to this study and be assigned to the test group or the control group. The subject will administer the first dose of assigned investigational product in the evening prior to the scheduled colonoscopy. Subject will take the second dose early in the morning of the colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who is informed and give a consent in voluntary
* Patients who is scheduled a colonoscopy
* BMI 19≤and<30

Exclusion Criteria:

* Patients who participate in other interventional study or had participated within 30 days before screening
* Pregnant or breast-feeding women who do not want to stop breast-feeding
* Women of childbearing potential who do not agree with appropriate contraception during this study
* Patients who had experienced any hypersensitivity study drug or ingredient
* Uncontrolled hypertension
* Arrhythmia with clinically significant findings from EKG
* Congestive heart failure; NYHA functional class III or IV; unstable coronary artery disease; myocardiac infarction history within 6 months
* Uncontrolled diabetes
* Active infection except acute upper respiratory infection or local skin infection; Fever (38 °C and higher) within 1 week before study administration
* HIV infection and/or chronic hepatitis B or C
* Patients who has a difficulty to participate because of severe nausea or vomiting
* Suspected or confirmed inflammatory bowel disease, toxic colon or toxic megacolon, or gastrointestinal obstruction or perforation; visible bleeding in colon
* History of colon surgery and abdominal surgery within 6 month; need an emergency surgery
* Colonoscopy for the following use: treatment of bleeding from such lesions as vascular malformation, ulceration, neoplasia, and polypectomy site (e.g.,electrocoagulation, heater probe, laser or injection therapy); foreign body removal; decompression of acute nontoxic megacolon or sigmoid volvulus; balloon dilation of stenotic lesions (e.g., anastomotic strictures); palliative treatment of stenosing or bleeding neoplasms (e.g., laser, electrocoagulation, stenting)
* Fluid or electrolyte (Na, K, Ca, Mg, chloride, bicarbonate) disturbance
* Severe dehydration risk (e.g., rhabdomyolysis, ascites)
* History of hypersensitivity of drug or others
* Alcohol or drug abuse within 6 months
* Clinically significant underlying disease or medical history at investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Successful cleansing rate | Two days (from day of first dosing to day of colonoscopy)
  %Patient with HCS-graded A or B

SECONDARY OUTCOMES:
Overall cleansing rate | Two days (from day of first dosing to day of colonoscopy)
  %Patient with each HCS-grade (A, B, C, D)
Mean segmental cleansing score | Two days (from day of first dosing to day of colonoscopy)
  Mean HCS-grade in each segment (5 Segments: Rectum, Sigmoid colon, Descending colon, Transverse colon, Ascending colon/cecum)
Mean cecal intubation time | Two days (from day of first dosing to day of colonoscopy)
Mean colonoscopy withdrawal time | Two days (from day of first dosing to day of colonoscopy)
Treatment compliance | Two days (from day of first dosing to day of colonoscopy)
  %Patient who have completed taking the investigational products
Patient satisfaction | Two days (from day of first dosing to day of colonoscopy)
  Patient questionnaire about any patient discomfort related to investigational products
Polyp detection rate | Two days (from day of first dosing to day of colonoscopy)

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Chonnam National University Hospital, Gwangju
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyunghee University Hospital, Seoul
  - Seoul National University Hospital, Seoul